CLINICAL TRIAL: NCT06942091
Title: Impact of Traumatic Brain Injury on Concomitant Blunt Hollow Organ Injuries: A Retrospective Analysis of a Cohort of Blunt Bowel Mesenteric Injuries
Brief Title: Impact of Traumatic Brain Injury on Hemodynamic Instability in Patients With Blunt Bowel and Mesenteric Injuries
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shih-Chiang Hung, Attending Physician, Chang Gung Memorial Hospital
Other Study IDs: 201902275B0
Record Dates: First submitted 2025-04-13; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Brain Injury; Blunt Abdominal Trauma; Hemodynamic Instability; Shock; Massive Transfusion
MeSH Terms: conditions — Brain Injuries, Traumatic; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TBI Group/non-TBI Group: TBI Group: Patients with blunt bowel and mesenteric injury (BBMI) with concomitant traumatic brain injury (TBI) Non-TBI Group: Patients with blunt bowel and mesenteric injury (BBMI) without TBI
  Interventions: Other: Traumatic Brain Injury (TBI)

INTERVENTIONS:
Other: Traumatic Brain Injury (TBI) — Presence of TBI identified by intracerebral hemorrhage on brain computed tomography (CT) at emergency department; not actively assigned by investigators but used to stratify comparison groups.

SUMMARY:
This retrospective cohort study aims to evaluate the impact of traumatic brain injury (TBI) on hemodynamic status in trauma patients with surgically confirmed blunt bowel and mesenteric injuries (BBMI). A total of 169 adult patients treated at a Level I trauma center between 2009 and 2023 were analyzed and stratified based on the presence or absence of concomitant TBI. Clinical parameters such as shock, massive transfusion, transfusion requirements, morbidity, and mortality were compared. The study investigates whether TBI is an independent risk factor for acute hemodynamic instability in BBMI patients, with the goal of improving trauma care strategies and understanding the systemic effects of TBI, particularly through the lens of the brain-gut axis.

DETAILED DESCRIPTION:
Patients Population We retrospectively reviewed patients with BBMI admitted to emergency department (ED) of Kaohsiung Chang Gung Memorial Hospital during the 15-year period January 1, 2009 to December 31, 2023 from the electronic medical record. Adult patients (age > 16 years of age) receiving therapeutic laparotomy for proven of BBMI were included in the study. Patient with isolated stomach, duodenal, or rectal injuries was excluded. Among these enrolled patients receiving brain computed tomography (CT) obtained at the ED, showing any type of intracerebral hemorrhage was defined as TBI (AIS ≥3). Patients were grouped according to the presence of intracerebral hemorrhage in the positive TBI versus negative TBI group. The two groups were compared, and associated injuries were assessed for their ability to predict the risk factors of presence of shock and receiving massive transfusion (MT), indicating of hemodynamic instability.

Study settings All trauma patients were treated according to the Advanced Trauma Life Support upon arrival to ED. Injury severity was calculated as Injury Severity Score (ISS) and New Injury Severity Score (NISS) based on the Abbreviated Injury Score (AIS) score[19]. Trauma Score Injury Severity Score (TRISS) was used for prediction of prognosis. Laboratory data including leukocyte and hemoglobin were measured from samples obtained at ED. The demographic data, injury mechanism, vital signs, and Glasgow Coma Scores up on arrival to ED were recorded. Regarding the clinical presentation, the procedures including receiving endotracheal tube intubation, and tube thoracostomy at the ED, and presence of shock episode which was defined as systolic blood pressure < 90 mmHg were recorded. The incidence of need of transfusion at ED and MT defined as receiving more than 10 units packed red blood cells (RBC) within 24 hours was recorded. The amount of transfused Pack RBC or fresh frozen plasma (FFP) at the ED, operative room (OR) or within the initial 24 hours was recorded as well. Operative findings including the incidence of isolated small bowel injury (defined as only small bowel injury including ischemia, rupture, serosa injury, or hematoma), isolated colon injury (defined as only colon injury), isolated mesentery injury (defined as only mesenteric injury), combined injury (defined as either small bowel or colon injury concomitant with mesenteric injury), and operative blood loss were recorded. The outcomes including morbidity, mortality regarding 24 hour mortality, bowel-related or exsanguinations related, and length of stay regarding intensive care unit (ICU) and hospitalization were recorded.

The development of post injury complications including sepsis, pneumonia, septic shock, unplanned ventilator, intraabdominal abscess, postoperative leakage, coagulopathy, acute renal failure, acidosis, urinary tract infection, stroke, pulmonary embolism, acute respiratory distress syndrome, pleural effusion, enterocutaneous fistula, wound infection, abdomen compartment syndrome, tracheostomy, extracorporeal membrane oxygenation (ECMO), return to the operating room, and hemodialysis, intestinal obstruction was registered and defined as morbidity.

Statistics The data were analyzed using IBM SPSS Statistics for Windows, version 20.0 (IBM Corp., Armonk, NY, USA). Continuous variables were reported as medians and interquartile ranges. Considering the potential impact of a small sample size on our statistical analysis, we treated the data as non-normally distributed. The Mann-Whitney U test was therefore employed to analyze these continuous variables. We used logistic regression to evaluate the independent impact of TBI on presence of shock and receiving MT in BBMI patients while controlling for age, sex and associated injuries. Given that patients had varying degrees and different associated injuries, we considered the associated injuries as the possible confounders instead of the ISS due to its nonspecific nature and inability to differentiate injury patterns. To analyze the temporal relationship of TBI between morbidity and mortality, Kaplan-Meier analysis was utilized, and the log-rank test was applied to compare the morbidity and mortality curves between the TBI(+) and TBI(-) groups. The threshold for statistical significance was set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >16 years
* Patients with surgically confirmed blunt bowel and/or mesenteric injuries (BBMI)
* Underwent therapeutic laparotomy
* Complete emergency department and operative records available

Exclusion Criteria:

* Isolated gastric, duodenal, or rectal injuries
* Pediatric patients (<16 years)
* Incomplete or missing clinical records
* Penetrating trauma
* Patients who did not undergo surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult trauma patients underwent surgically confirmed blunt bowel and mesenteric injuries.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Presence of Shock | At Emergency Department (initial presentation)
  Proportion of BBMI patients who experienced shock, defined as systolic blood pressure < 90 mmHg at the emergency department.
Need for Massive Transfusion | Within 24 hours of hospital admission
  Proportion of BBMI patients who received more than 10 units of packed red blood cells within 24 hours after arrival.

SECONDARY OUTCOMES:
Amount of Transfusion Administered | Within 24 hours of hospital admission
  Total number of packed red blood cell (PRBC) and fresh frozen plasma (FFP) units transfused within 24 hours.
In-hospital Morbidity | Through hospital discharge, a median length of 17 days
  Proportion of patients developing at least one complication such as pneumonia, coagulopathy, acidosis, urinary tract infection, tracheostomy, etc.
In-hospital Mortality | Up to hospital discharge, a median length of 17 days
  All-cause mortality occurring during the index hospitalization.
ICU Length of Stay | Through ICU stay during index hospitalization, a median length of 3 days
  Duration of stay in the intensive care unit (ICU) in days.